CLINICAL TRIAL: NCT03548519
Title: Innovative Attention Training to Achieve Stable Remission in Depression: A Randomized Controlled Trial Study
Brief Title: Online Contingent Attention Training (OCAT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to technical reasons
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC/2018/0509
Record Dates: First submitted 2018-05-15; First posted 2018-06-07 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Major Depression in Remission

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Training (Experimental): OCAT-only: An attention training, consisting of 10 sessions of ±12 minutes each (during an intervention period of two weeks), will be administered. The training task is a positively directed Scrambled Sentences Test (SST) with mouse-gaze contingent feedback.
  Interventions: Behavioral: OCAT-only
- Active placebo training (Active Comparator): OCAT-sham: An active placebo training, consisting of 10 sessions of ±12 minutes each (during an intervention period of two weeks), will be administered. The training task is an undirected Scrambled Sentences Test (SST) with mouse-gaze contingent feedback.
  Interventions: Behavioral: OCAT-sham
- PSE and Attention Training (Experimental): OCAT-combo: An online PSE session prior to an attention training, consisting of 10 sessions of ±12 minutes each (during an intervention period of two weeks), will be administered. Content of the PSE will focus on how adaptive functions of automatic and controlled processes may become maladaptive when used inappropriately or excessively. The training task is a positively directed Scrambled Sentences Test (SST) with mouse-gaze contingent feedback.
  Interventions: Behavioral: OCAT-combo

INTERVENTIONS:
Behavioral: OCAT-only — online-contingent Attention Training without prior psychoeducation
  Arms: Attention Training
Behavioral: OCAT-sham — Placebo version of Online contingent Attention Training without prior psychoeducation
  Arms: Active placebo training
Behavioral: OCAT-combo — Online contingent Attention Training with prior psychoeducation
  Arms: PSE and Attention Training

SUMMARY:
This study evaluates the effectiveness of a smartphone-delivered attention control training as a preventive intervention for remitted depressed patients. Additionally, the investigators aim to increase the effect of this CBM-intervention by adding a psychoeducation module (CBT-intervention). To test this aim, participants will be randomly assigned to one of three conditions: (1) an experimental training condition with prior psychoeducation, (2) an experimental training condition without prior psychoeducation, or (3) a placebo training condition serving as an active control condition.

DETAILED DESCRIPTION:
According to different theories and empirical research, attention control for external information and cognitive control for internal information play a causal role in cognitive emotion regulation ability, a critically important factor in determining resilience. Recent studies regarding the more specific interplay among these mechanisms in depression highlight the importance of considering attention control in treating impaired emotion regulation processes. These studies tested an interactive attention control training, in which people learned to disentangle scrambled sentences ("life is my party a mess") in a positive way ("my life is a party") by receiving eye tracking-based feedback on attention for positive ("party") vs. negative information ("mess"). Results indicated that participants were better able to reinterpret negative pictures in a positive way. Moreover, reactive attentional and cognitive control (i.e., when actually being confronted with a challenging task or stressor) seem to be influenced by perceived control or expectancy regarding the ability to cope with future stressors (i.e., in anticipation of a challenging task or stressor). More specifically, low perceived control and negative expectation bias with respect to future emotion regulation ability have been shown to result in an increased need for actual control and decreased emotion regulation abilities when actually being confronted with stressors. Based on these findings, it could be assumed that the effects of attention control training - targeting actual controlled emotion regulation processes - may be improved by adding techniques that influence perceived control/expectancy of emotion regulation ability (e.g., psychoeducation).

In the current study, the investigators aim to investigate whether an online based variant of the eye-gaze contingent attention training could be a promising intervention for relapse prevention in people vulnerable to depression. More specifically, the main aim is to explore whether an online-delivered attention control training can improve depressive symptoms and cognitive emotion regulation ability (e.g., reappraisal ability), thereby increasing resilience in the face of stress, in a RMD (remitted depressed) sample. In addition, it will be explored whether prior psychoeducation may increase this effect.

In each condition, a smartphone training, consisting of 10 sessions of about 12 minutes each, will be administered to remitted depressed participants. The experimental condition will receive an attention training with gaze contingent feedback (OCAT), comprising an undirected interpretation task (instruction to unscramble as quickly as possible) as a baseline phase, followed by a positively directed interpretation task (instruction to unscramble always positive self-statements) as a modification phase (OCAT-only condition). The active placebo training will only receive the undirected interpretation task (modification phase identical to baseline phase) without mouse-gaze contingent feedback (OCAT-sham condition). Furthermore, an additional condition will combine the experimental training with a new psychoeducation session (OCAT-combo condition). This psychoeducation will focus on the role of attention processes in generating emotions. As the training tasks, this PSE-session will be self-administered and delivered in a computer-based format, including interactive graphics and video-recordings.

Before (pre-test) and after the intervention (post-test), selective attention bias and emotion regulation will be measured to investigate transfer effects of training. Also, depressive symptomatology and related variables will be assessed at pre- and post-test, as well as at follow-up, 3 and 6 months after the training.

ELIGIBILITY:
Inclusion Criteria:

* History of ≥ 1 depressive episodes (major or bipolar)
* Currently in stable full or partial remission (≥ 3 months)
* Being in possession of a recent computer (needed to install the training software)

Exclusion Criteria:

* Major depressive disorder (current or less than 3 months in remission)
* Bipolar disorder (current or less than 3 months in remission)
* Psychotic disorder (current and/or previous)
* Neurological impairments (current and/or previous)
* Excessive substance abuse (current and/or previous)
* Ongoing psychotherapeutic treatment (maintenance treatment is allowed, but with a frequency of less than once every three weeks)
* Use of antidepressant medication is allowed if kept at a constant level
* Not being in possession of a recent computer (needed to install the training software)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in depression, anxiety, and stress | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the 21-item version of the Depression, Anxiety, and Stress Scales (DASS-21)
Change in rumination | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the Ruminative Response Scale (RRS). This 22-item questionnaire provides a total rumination score (range: 22 - 88), as well as Brooding and Reflection subscale scores (range: 5 - 20). Brooding is characterized by a passive style of moody pondering and is the most maladaptive form of depressive rumination. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Change in attentional bias | Pre-test, Post-test (immediately after the two week intervention period)
  Measured by an emotional dot-probe task
Change in reappraisal | Pre-test, Post-test (immediately after the two week intervention period)
  Measured by the emotion regulation task: Average of two blind raters' scores of participants' reappraisal descriptions on a 5-point scale (0-No Description, 1-Not at all, 2-A little, 3-Good, 4-Very good) on participants' ability to reinterpret negative scenes (separately for the pre- and post-test emotion regulation tasks)
Change in negative emotions (after reappraisal) | Pre-test, Post-test (immediately after the two week intervention period)
  Measured by the emotion regulation task: Average of negative mood ratings after using reappraisal
Change in (mal-)adaptive cognitive emotion regulation strategies | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the Cognitive Emotion Regulation Questionnaire (CERQ)
Change in maladaptive cognitive emotion regulation strategies: State rumination | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the Brief State Rumination Inventory (BSRI)
Change in general functioning: Quality of life | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the depression-specific 34-item (range: 0 - 34) Quality of Life in Depression Scale (QLDS). The QLDS consists of dichotomous response questions, with the response being either True/Not True or Yes/No. It is scored binomially (0-1) and high scores on the QLDS indicate a lower quality of life.
Change in general functioning: Remission from depression | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the 41-item Remission of Depression Questionnaire (RDQ) for which a high score is indicative for more psychopathology (range: 0 - 82).
Change in general functioning: Resilience | Pre-test, Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the Connor-Davidson Resilience Scale (CD-RISC). The CD-RISC comprises of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience.
Treatment Credibility and Expectancy | Pre-test, Post-test (immediately after the two week intervention period)
  Measured by the Credibility/Expectancy Questionnaire (CEQ)
Change in motivation-related variables | Post-test (immediately after the two week intervention period), Follow-up (3 and 6 months)
  Measured by the Intrinsic Motivation Inventory (IMI). Subscales: Interest/Enjoyment, Perceived Competence, Effort/Importance, Pressure/Tension, Value/Usefulness

OTHER OUTCOMES:
User engagement | Post-test (immediately after the two week intervention period)
  Measured by the 31-item User Engagement Scale (UES). The UES comprises 6 subscales of engagement: Focused attention (FA; 7 items); Perceived usability (PU; 8 items), Aesthetic appeal (AE; 5 items), Endurability (EN; 5 items), Novelty (NO; 3 items), and Felt involvement (FI; 3 items). Scale scores are calculated for each participant by summing scores for the items in each of the six subscales and dividing by the number of items. To calculate an overall engagement score, the average of each of the six subscales of the UES long form should be summed. Higher scores indicate higher engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Koster, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez A, Everaert J, Koster EH. Attention training through gaze-contingent feedback: Effects on reappraisal and negative emotions. Emotion. 2016 Oct;16(7):1074-85. doi: 10.1037/emo0000198. Epub 2016 Jun 20. PMID 27322115
- [Background] Vanderhasselt MA, De Raedt R, De Paepe A, Aarts K, Otte G, Van Dorpe J, Pourtois G. Abnormal proactive and reactive cognitive control during conflict processing in major depression. J Abnorm Psychol. 2014 Feb;123(1):68-80. doi: 10.1037/a0035816. PMID 24661161